CLINICAL TRIAL: NCT06972160
Title: Interventions to Increase Adherence to Colorectal Cancer Screening in Barcelos/Esposende: a Randomized Clinical Trial
Brief Title: Intervention Project to Increase Adherence to Colorectal Cancer Screening in Barcelos/Esposende
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Local Health Unit Barcelos/Esposende, Public Health Unit (Other Government)
Collaborators: Instituto de Saude Publica da Universidade do Porto (Other)
Responsible Party: Principal Investigator, David Nascimento Moreira, Public Health Medical Doctor, Local Health Authority, Instituto de Saude Publica da Universidade do Porto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: Rede+Rastreio-Cancro
Record Dates: First submitted 2025-04-16; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Colon and Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional Group (Experimental): The interventional group will be subjected to interventions to increase the adherence to screening, including text messages via phone as well as phone calls.
  Interventions: Other: Arm1: intervention 1 (SMS+call)
- Control group (Placebo Comparator): The control group will not be subjected to any interventions to increase the adherence to screening.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Arm1: intervention 1 (SMS+call) — The intervention will consist in two text messages (one and two weeks after received the screening test, respectively), an automated non-human call or a call made by the administrative assistant (three weeks after received the screening test), and a phone call made by a physician (four weeks after received the screening test)
  Arms: Interventional Group
Other: Control group — The control group will not be subjected to any interventions to increase the adherence to screening.
  Arms: Control group

SUMMARY:
An experimental study through a randomized clinical trial, without blinding (for participants and the research team), with a control group (not subject to intervention) and an intervention group (subject to two text messages, an automated non-human call or a call made by the administrative assistant, and a phone call made by a physician).

ELIGIBILITY:
Inclusion Criteria:

Participants must be registered in the ULS of

Barcelos/Esposende and meet the following criteria:

1. Age between 50 and 74 years.
2. No symptoms such as weight loss in the last 6 months or gastrointestinal symptoms.
3. No prior diagnosis of CRC.
4. No diagnosis of inflammatory bowel disease (ulcerative colitis or Crohn's disease).
5. No family history of CRC in first- and second-degree relatives diagnosed before age 60.
6. No prior fecal occult blood test (FOBT) in the 11 months before receiving the collection kit or no prior sigmoidoscopy or colonoscopy in the last 24 months.

Exclusion Criteria:

1. Participants who did not receive the screening kit at home.
2. Participants without a phone number.
3. Participants who do not answer the phone or refuse to participate in the study.
4. Participants unable to consent or perform the screening due to physical, mental, or other conditions that seriously impair comprehension.

Ages: 49 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1038 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Adherence to colon and rectal screening [Time Frame: 6 weeks] | From April 2025 to June 2025 (6 weeks)
  Increase in adherence to colon and rectal screening
  Proportion/cumulative proportion of patients who performed colon and rectal cancer screening among those who were invited to undergo it, after step 1 (SMS1), step 2 (SMS2), step 3 (administrative call) and step 4 (medical doctor call)

CONTACTS AND LOCATIONS:
Locations (1):
- Public Health Unit Barcelos/Esposende, Porto, Portugal

IPD SHARING:
Plan to Share IPD: Undecided
We plan to share de-identified individual participant data (IPD) that underlie the results reported in this study, including text, tables, and figures. The data will be made available beginning six months after publication and will remain accessible for a period of five years. Access will be granted to researchers who submit a methodologically sound proposal, subject to approval by the study team. Along with the IPD, supporting documents such as the study protocol, statistical analysis plan, and informed consent form will also be available. Requests for data access should be directed to Marina Pinheiro, MD, PhD email: mpinheiro@icbas.up.pt.